CLINICAL TRIAL: NCT04108299
Title: Feasibility of a Family-oriented mHealth Intervention for Chinese Americans With Type 2 Diabetes
Brief Title: Family Intervention for Chinese Americans With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 19-01275
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes
Keywords: Chinese Americans
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-list Control (Placebo Comparator): Standard of care
  Interventions: Behavioral: Wait-list control group
- SMS Intervention (Experimental): The SMS group will receive brief lifestyle counseling videos via SMS links. At the end of the study, the wait-list control group will be provided the opportunity to receive the counseling videos.
  Interventions: Behavioral: SMS intervention

INTERVENTIONS:
Behavioral: Wait-list control group — For patient participants, they will continue to receive the standard of usual care for their T2D at the CBWCHC during the course of our study. For family/friend participants, they will continue to receive their routine care with their own doctors during the study. At the end of the study, the wait-list control group (both patient and family/friend participants) will be provided the opportunity to receive the counseling videos delivered to them via SMS links.
  Arms: Wait-list Control
Behavioral: SMS intervention — 2-3 SMS-based diabetes videos will be sent to patients each week for 12 weeks (each video within 10 minutes in duration) to both patients and their family members. Patients and their family members will receive the same intervention videos, including basic information about T2D, importance of diabetes self-management at home, behavioral techniques, and family-oriented sessions. BrainShark will be used to determine whether participants view these,videos. For participants who miss 3 consecutive videos, the study team will follow-up with a phone call to identify barriers to watching the video and remind them to review the video.
  Arms: SMS Intervention

SUMMARY:
The goal of this pilot study is to examine the feasibility and acceptability of a family-oriented SMS intervention in 30 Chinese Americans with T2D and their family members. Participants will be randomized to one of 2 arms (n=15 each): 1) wait-list control and 2) SMS intervention. Both groups will continue to receive standard of care treatment for their T2D. The SMS group will receive brief lifestyle counseling videos via SMS links. At the end of the study, the wait-list control group will be provided the opportunity to receive the counseling videos.

DETAILED DESCRIPTION:
Chinese Americans are one of the fastest growing immigrant groups in the US, who suffer disproportionately high type 2 diabetes (T2D) burden and have poorly controlled T2D. Given the high economic and societal burden of T2D and rapid population growth in Chinese Americans, there is an urgent need for research to develop effective interventions to address T2D burden in this population. Recent evidence suggests the importance of involving and empowering family members in diabetes intervention and calls for family intervention. A mobile health approach such as short message service (SMS) might be a promising way to deliver such family-oriented interventions to the target population given prior studies suggests that Chinese Americans often report challenges to attend in-person lifestyle counseling because of long working hours and lack of sick time from work. A SMS-based intervention provides the flexibility of allowing them to view the intervention at a time and place convenient to them. This study will serve as the first step to explore an alternative approach for managing T2D in this group.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patient participants:

* self-identify as Chinese or Chinese American;
* be between the ages of 18 and 70,
* self-report a diagnosis of T2D;
* be willing to receive WeChat messages regarding T2D management,
* possess a smartphone or be willing and able to use a study smartphone. If participants have their own smartphones, they are encouraged to use their own phones. For participants who do not have smartphones, the study will provide them
* has a family member or friend be willing to participate in the study to learn about T2D to better support them

Inclusion criteria for family/friend participants: family/friend participants must

* be between 18-70 years old,
* be willing to receive WeChat messages regarding T2D management
* possess a smartphone or be willing and able to use a study smartphone. If participants have their own smartphones, they are encouraged to use their own phones. For participants who do not have smartphones, the study will provide them

Exclusion Criteria:

Exclusion criteria for both patient and family/friend participants:

* unable or unwilling to provide informed consent;
* unable to participate meaningfully in the intervention (e.g., uncorrected sight and hearing impairment);
* unwilling to accept randomization assignment;
* pregnant, plans to becomes pregnant in the next 6 months, or who become pregnant during the study, or
* breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hu, PhD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Requests should be directed to lu.hu@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Wait-list Control - Patients; Wait-list Control - Family/Friend; SMS Intervention - Family/Friend: Standard of care
  Wait-list control group: For patient participants, they will continue to receive the standard of usual care for their T2D at the CBWCHC during the course of our study. For family/friend participants, they will continue to receive their routine care with their own doctors during the study. At the end of the study, the wait-list control group (both patient and family/friend participants) will be provided the opportunity to receive the counseling videos delivered to them via SMS links.
- SMS Intervention - Patients: The SMS group will receive brief lifestyle counseling videos via SMS links. At the end of the study, the wait-list control group will be provided the opportunity to receive the counseling videos.
  SMS intervention: 2-3 SMS-based diabetes videos will be sent to patients each week for 12 weeks (each video within 10 minutes in duration) to both patients and their family members. Patients and their family members will receive the same intervention videos, including basic information about T2D, importance of diabetes self-management at home, behavioral techniques, and family-oriented sessions. BrainShark will be used to determine whether participants view these,videos. For participants who miss 3 consecutive videos, the study team will follow-up with a phone call to identify barriers to watching the video and remind them to review the video.
Period: Overall Study
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Started | 12 | 11 | 12 | 11
Completed | 10 | 10 | 10 | 10
Not Completed | 2 | 1 | 2 | 1
Not completed — Not interested in participating | 2 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend | Total
Number analyzed (Participants) | 12 | 11 | 12 | 11 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.92 (7.62) | 55.45 (11.45) | 61.7 (5.98) | 48.18 (11.04) | 55.42 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 7 | 23
  Male | 6 | 6 | 7 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 12 | 11 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 11 | 12 | 11 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 12 | 11 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Videos Watched by Participants
Description: Measure of SMS intervention feasibility.
Time Frame: Up to Month 6
Population: Population comprises 10 participants and 10 family members/friends in the SMS Intervention Group. Participants in the Wait-list Control group were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of videos watched
Arm/Group | SMS Intervention
Number analyzed (Participants) | 20
Percentage of videos watched | 76.8 (7)

2. Primary Outcome: Satisfaction Questionnaire Score
Description: 1-item assessment of satisfaction with the SMS intervention. The item is rated on a scale from 0 (not at all satisfied) to 10 (totally satisfied). The total score is the numerical response; higher scores indicate greater satisfaction.
Time Frame: Month 6
Population: Participants in the Wait-List Control arm were not assessed for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SMS Intervention - Patients | SMS Intervention - Family/Friend
Number analyzed (Participants) | 10 | 10
score on a scale | 9.4 (1) | 10 (0)

3. Secondary Outcome: Change in HbA1c Level
Description: Participants receive HbA1c blood test at their doctors' office every 3-6 months; HbA1c testing results will be abstracted from the medical record at the participant's health care facility.
Time Frame: Baseline, Month 6
Population: Change in HbA1c level was not assessed in family/friend participants.
Measure: Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients
Number analyzed (Participants) | 12 | 11
percentage of glycosylated hemoglobin | -0.88 [-1.81 to 0.05] | -1.23 [-2.21 to -0.24]

4. Secondary Outcome: Change in Body Weight
Description: Body weight in pounds (lbs).
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: lbs
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
lbs | -4.75 [-17.68 to 8.18] | -11.68 [-24.71 to 1.35] | -4.88 [-29.06 to 19.30] | -2.59 [-25.24 to 20.06]

5. Secondary Outcome: Change in Diabetes Management Self-Efficacy Scale (DMSES) Score
Description: The DMSES is an 8-item assessment asking participants to rate their confidence level in performing diabetes-specific self-management behaviors, using a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident). The total score is the sum of responses and ranges from 8 to 80; higher scores indicate greater self-efficacy. An increase in scores indicates self-efficacy improved during the observational period.
Time Frame: Baseline, Month 6
Population: Change in DMSES Score was not assessed in family/friend participants.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients
Number analyzed (Participants) | 12 | 11
Score on a scale | 0.43 [-0.61 to 1.46] | 0.38 [-0.68 to 1.44]

6. Secondary Outcome: Change in Summary of Diabetes Self-Care Activities (SDSCA) Score
Description: The SDSCA is a 13-item assessment of participants' adherence to diabetes self-management behaviors. This scale consists of 13 items and asks participate to describe their diabetes self-care activities over the past 7 days. The total score is the sum of responses and ranges from 0 to 91; higher scores indicate greater adherence to self-management behaviors. An increase in scores indicates adherence improved during the observational period.
Time Frame: Baseline, Month 6
Population: Change in SDSCA score was not assessed in family/friend participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients
Number analyzed (Participants) | 12 | 11
score on a scale | 7.15 [-0.26 to 14.57] | 10.05 [2.56 to 17.53]

7. Secondary Outcome: Change in Diabetes Knowledge Test Scores
Description: 11-item questionnaire assessing diabetes knowledge. The total score is the number of correct responses and ranges from 0-11.
Time Frame: Baseline, Month 6
Population: Patient participants were not assessed for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11
score on a scale | 0.14 [0.00 to 0.29] | 0.24 [0.11 to 0.37]

8. Secondary Outcome: Change in International Physical Activity Questionnaire (IPAQ)-Short Version MET Score
Description: The IPAQ calculates each participant's metabolic equivalent (MET) score by asking participants the days and minutes exercised in three categories of intensity (vigorous, moderate, and walking) during the previous one week. One metabolic equivalent (MET) is defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min. Higher MET scores indicate higher levels of physical activity. An increase in scores indicates physical activity increased during the observational period.
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Metabolic equivalent (MET)
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
Metabolic equivalent (MET) | 1656.37 [-735.69 to 4048.44] | 1076.7 [-1340.2 to 3493.59] | 329.71 [-986.25 to 1645.67] | 765.84 [-418.10 to 1949.79]

9. Secondary Outcome: Change in Mediterranean Dietary Screener (MEDAS) - Fruit Score
Description: The MEDAS contains 6 items and asks respondents about the types of food they consumed in the past 30 days: 1) fruits, 2) vegetables, 3) refined grains, 4) whole wheat, 5) sugary drinks, and 6) starchy foods. For each type of food, respondents estimate the amount (in cups) of the food they have eaten each day over the past 30 days. Higher scores indicate higher consumption of the food group analyzed.
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: cups
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
cups | 0.07 [-0.37 to 0.51] | 0.08 [-0.36 to 0.52] | 1.03 [0.43 to 1.62] | -0.18 [-0.71 to 0.36]

10. Secondary Outcome: Change in Mediterranean Dietary Screener (MEDAS) - Vegetable Score
Description: as for outcome 9
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: cups
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
cups | 0.57 [0.00 to 1.15] | 0.41 [-0.17 to 0.99] | 1.18 [0.31 to 2.05] | -0.18 [-0.96 to 0.61]

11. Secondary Outcome: Change in Mediterranean Dietary Screener (MEDAS) - Refined Grains Score
Description: as for outcome 9
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: cups
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
cups | -0.31 [-0.70 to 0.07] | -0.09 [-0.48 to 0.29] | -0.39 [-0.95 to 0.17] | -0.68 [-1.18 to -0.17]

12. Secondary Outcome: Change in Mediterranean Dietary Screener (MEDAS) - Whole Wheat Score
Description: as for outcome 9
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: cups
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
cups | -0.32 [-0.91 to 0.27] | 0.16 [-0.44 to 0.77] | 0.44 [0.15 to 0.73] | -0.09 [-0.36 to 0.17]

13. Secondary Outcome: Change in Mediterranean Dietary Screener (MEDAS) - Sugary Drinks Score
Description: as for outcome 9
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: cups
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
cups | -0.22 [-0.48 to 0.04] | -0.31 [-0.58 to -0.04] | -0.19 [-0.52 to 0.14] | -0.23 [-0.53 to 0.08]

14. Secondary Outcome: Change in Mediterranean Dietary Screener (MEDAS) - Starchy Score
Description: as for outcome 9
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: cups
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
cups | 0 [-0.20 to 0.21] | -0.07 [-0.28 to 0.14] | -0.03 [-0.21 to 0.16] | -0.07 [-0.24 to 0.09]

15. Secondary Outcome: Change in Diabetes-Specific Support Score
Description: Participants were asked about diabetes-specific support, such as medication taking, healthy diet, physical activity, blood sugar monitoring, stress management, and diabetes management. Higher scores indicate better support. The total score ranges from 4-80; higher scores indicate greater levels of specific.
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
score on a scale | 6.92 [-0.73 to 14.58] | 3.15 [-4.70 to 11.00] | 9.22 [-0.72 to 19.16] | 9.12 [-0.12 to 18.35]

16. Secondary Outcome: Change in the Patient Reported Outcome Measurement Information System (PROMIS) Emotional Support Short Form v2.0 Score
Description: 4-item assessment of the availability of others with whom they could talk and feel appreciated. The total score ranges from 4 - 20; higher scores indicate greater support.
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
Number analyzed (Participants) | 12 | 11 | 12 | 11
score on a scale | 0.64 [0.08 to 1.19] | 0.63 [0.07 to 1.19] | 0.7 [0.50 to 1.91] | 1.2 [0.06 to 1.34]

17. Secondary Outcome: Change in Diabetes Distress Scale Score
Description: The Diabetes Distress Scale consists of 17 items and asks respondents to describe the diabetes-related distress experienced within the past month, including emotional distress, physician-related distress, regimen-related distress, and interpersonal distress. The items are scored on a 6- point Likert scale, ranging from 1 (not a problem) to 6 (a very serious problem). The total score is the sum of responses and ranges from 17 to 102, with higher scores indicating higher levels of diabetes distress.
Time Frame: Baseline, Month 6
Population: Family/friend participants were not assessed for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients
Number analyzed (Participants) | 12 | 11
score on a scale | -0.67 [-1.35 to 0.01] | -0.5 [-1.20 to 0.19]

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Wait-list Control - Patients | SMS Intervention - Patients | Wait-list Control - Family/Friend | SMS Intervention - Family/Friend
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT04108299/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT04108299/ICF_000.pdf